CLINICAL TRIAL: NCT00963027
Title: An Evaluation of Single Dose UT-15C SR (Treprostinil Diethanolamine) Pharmacokinetics Following Repeated Dosing With the Proton Pump Inhibitor Esomeprazole in Healthy Adult Volunteers
Brief Title: Effect of Esomeprazole on the Pharmacokinetics of Oral Treprostinil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Allison Pecha, United Therapeutics, Corp.
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-116
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Hypertension, Pulmonary; Pulmonary Arterial Hypertension
Keywords: Hypertension, Pulmonary; Treprostinil; Pharmacokinetics; Treprostinil Diethanolamine; Pulmonary Arterial Hypertension; Esomeprazole
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treprostinil diethanolamine — Subjects will each receive a single 1 mg sustained release tablet of treprostinil diethanolamine by mouth immediately following breakfast before and after repeated daily dosing with esomeprazole.
  Other Names: UT-15C; UT-15C SR; Oral treprostinil
Drug: Esomeprazole — Each subject will receive a single 40 mg capsule of esomeprazole by mouth in the morning for seven days.
  Other Names: Nexium

SUMMARY:
The purpose of this study is to evaluate the effect of esomeprazole, a proton pump inhibitor, on treprostinil pharmacokinetics.

DETAILED DESCRIPTION:
This open-label study will evaluate the effect of esomeprazole, a proton pump inhibitor, on treprostinil pharmacokinetics following a single 1 mg oral dose of UT-15C SR in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy and between the ages of 18 and 55 years, inclusive, at Screening.
* Female subjects must weigh between 45 and 100 kg, inclusive, with a BMI between 19.0-29.9 kg/m2, inclusive at Screening. Male subjects must weigh between 50 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening.
* Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening.

Exclusion Criteria:

* Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
* Subject has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
* Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Treprostinil pharmacokinetics in healthy volunteers following a single oral dose of a 1 mg treprostinil diethanolamine sustained release tablet before and after repeated dosing with esomeprazole. | Within 10 minutes prior to through 36 hours post treprostinil diethanolamine dosing
Adverse event monitoring | Time Frame: From the first dose of treprostinil diethanolamine through study end (Study Day 9/10)

SECONDARY OUTCOMES:
Clinical laboratories | Study Days 0 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Laurent, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States